CLINICAL TRIAL: NCT04814186
Title: A Study to Characterize the Safety and Efficacy of Tafamidis Once Daily in the Treatment of Transthyretin Amyloid Cardiomyopathy in Chinese Participants
Brief Title: A Study to Assess the Safety and Efficacy Of Tafamidis In Chinese Participants With Transthyretin Amyloid Cardiomyopathy (ATTR-CM)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B3461077
Record Dates: First submitted 2021-03-10; First posted 2021-03-24 (Actual); Results first posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-11

CONDITIONS: Transthyretin Amyloid Cardiomyopathy
Keywords: Tafamidis
MeSH Terms: interventions — tafamidis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Chinese participants treated with Tafamidis (Experimental): treatment group with tafamidis
  Interventions: Drug: Tafamidis

INTERVENTIONS:
Drug: Tafamidis — 61 mg, once daily, oral administration, for 12 months.
  Other Names: Vyndamax, Tafamidis free acid, PF 06291826

SUMMARY:
This is a national, multi-center, single-arm study, open-label to patients with symptomatic Transthyretin amyloid cardiomyopathy (ATTR-CM) who are tafamidis naïve. This study is to obtain safety, descriptive efficacy, Pharmacokinetics (PK) and Pharmacodynamics (PD) data for tafamidis orally once daily.

Subject eligibility for participation in the study will receive tafamidis once daily or 12 months following the assessment as the screening and baseline, month 1, 3, 6, 9 and 12 visits (or Early Study Discontinuation).

ELIGIBILITY:
Inclusion Criteria:

1. Subject has documented ATTR-CM.
2. For the reproductive criteria for male and female participants, please refer to relevant protocol sections.

Exclusion Criteria:

1. Other acute or chronic medical or psychiatric condition including recent or active suicidal ideation or behavior or laboratory abnormality, in the judgment of the investigator, would make the participant inappropriate for entry into this study.
2. Participants who have prior liver and/or heart transplant.
3. Participants with primary (light chain) or secondary amyloidosis.
4. Previous administration with an investigational drug within 30 days or 5 half lives preceding the first dose of study intervention used in this study (whichever is longer).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2021-07-22 (Actual); Primary Completion 2023-10-16 (Actual); Study Completion 2023-10-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (9):
- China (9):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science & Technology, Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Tian Z, Peng D, Ma W, Yan J, Wang J, Tang Y, Jin W, Liu Y, Jia C, Gao Y, Gong Y, Sun X, Chen N, Zhu S, Zhang S. Safety and Efficacy of Tafamidis in Chinese Patients with Transthyretin Amyloid Cardiomyopathy. Cardiol Ther. 2025 Sep;14(3):439-452. doi: 10.1007/s40119-025-00408-6. Epub 2025 May 23. PMID 40410537
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B3461077

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 53 participants were enrolled in this study.
Groups:
- All Participants: Participants received tafamidis free acid 61 milligrams (mg) once daily (QD). Participants were instructed to take the study intervention on a daily basis (up to a maximum of 1 year).
Period: Treatment Phase
Arm/Group | All Participants
Started | 53
Completed | 43
Not Completed | 10
Not completed — Adverse Event | 1
Not completed — Death | 6
Not completed — Withdrawal by Subject | 2
Not completed — Other | 1
Period: Follow-Up Phase
Arm/Group | All Participants
Started | 53
Completed | 44
Not Completed | 9
Not completed — Adverse Event | 1
Not completed — Death | 6
Not completed — Withdrawal by Subject | 1
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all enrolled participants who took at least 1 dose of tafamidis free acid 61 mg soft capsule.
Arm/Group | All Participants
Number analyzed (Participants) | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 36
  >=65 years | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 47
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 53

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With All-Causality Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. All AEs that started after the first dosing but before the last dose plus the lag time (28 days) were TEAEs. A serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience; persistent disability/incapacity; congenital anomaly/birth defect. A severe TEAE was an event that prevented normal everyday activities. Severe TEAEs were assessed by the investigator.
Time Frame: From first dose of study intervention on Day 1 (baseline) up to 28 days post the last dose of study intervention (up to a maximum of 393 days)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 53
Participants
  TEAEs | 45
  Treatment-Emergent SAEs | 21
  Severe TEAEs | 17
  TEAEs Leading to Death | 6
  Discontinuations From Study Due to TEAEs | 1
  Permanent Discontinuations From Study Intervention Due to TEAEs | 1
  Dosing Interruptions of the Study Intervention due to TEAEs | 3

2. Primary Outcome: Number of Participants With Treatment-Related TEAEs
Description: An AE was any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. All AEs that started after the first dosing but before the last dose plus the lag time (28 days) were TEAEs. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience; persistent disability/incapacity; congenital anomaly/birth defect. A severe TEAE was an event that prevented normal everyday activities. Severe TEAEs and treatment-related TEAEs were assessed by the investigator.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 53
Participants
  TEAEs | 3
  Treatment-Emergent SAEs | 0
  Severe TEAEs | 0
  TEAEs Leading to Death | 0
  Discontinuations From Study Due to TEAEs | 0
  Permanent Discontinuations From Study Intervention Due to TEAEs | 0
  Dosing Interruptions of the Study Intervention due to TEAEs | 1

3. Secondary Outcome: Change From Baseline (CFB) for Distance Walked During 6 Minute Walk Test (6MWT) at Months 6 and 12
Description: As a measure of functional capacity, the 6MWT measured the distance a participant could walk on a straight course in 6 minutes. 6MWT was conducted in accordance with guidelines established by the American Thoracic Society at Month 6 and Month 12 visits. Baseline was defined as the last measurement prior to first dose of study intervention.
Time Frame: Baseline, months 6 and 12
Population: Efficacy analysis set included all enrolled participants who took at least 1 dose of tafamidis free acid 61 mg soft capsule. Number of Participants Analyzed represents the total number of participants in the efficacy analysis set regardless of the type of outcome measures. Number Analyzed for each row represents the number of participants who had a reportable measurement of 6MWT at baseline, at Months 6 (for reporting CFB at Month 6) and 12 (for reporting CFB at Month 12).
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | All Participants
Number analyzed (Participants) | 53
Meters
  Month 6: number analyzed (Participants) | 34
  Month 6 | -19.3 (73.36)
  Month 12: number analyzed (Participants) | 26
  Month 12 | 1.5 (91.29)

4. Secondary Outcome: Change From Baseline for N Terminal Prohormone B Type Natriuretic Peptide (NT-proBNP) at Months 6 and 12
Description: Plasma NT-proBNP is a guideline-mandated biomarker in heart failure. Baseline was defined as the last measurement prior to the first dose of study treatment.
Time Frame: Baseline, months 6 and 12
Population: Efficacy analysis set included all enrolled participants who took at least 1 dose of tafamidis free acid 61 mg soft capsule. Number of Participants Analyzed represents the total number of participants in the efficacy analysis set regardless of the type of outcome measures. Number Analyzed for each row represents the number of participants who had a reportable measurement of NT-proBNP at baseline, at Months 6 (for reporting CFB at Month 6) and 12 (for reporting CFB at Month 12).
Measure: Mean (Standard Deviation); unit: Nanograms per liter (ng/L)
Arm/Group | All Participants
Number analyzed (Participants) | 53
Nanograms per liter (ng/L)
  Month 6: number analyzed (Participants) | 45
  Month 6 | 452.9 (2625.04)
  Month 12: number analyzed (Participants) | 40
  Month 12 | -422.2 (1581.82)

5. Secondary Outcome: Percentage of Responders in Transthyretin (TTR) Stabilization Post Dose at Months 1, 6, and 12
Description: Blood sample of approximate 10 mL was collected at baseline, Months 1, 6, and 12 visits for measurement of TTR and TTR tetramer concentrations. TTR concentration was obtained prior to urea denaturation and TTR tetramer concentration was obtained after urea denaturation. Month 1 visit occurred 1 month post Day 1 +/- 1 week, Month 6 visit occurred 6 months post Day 1 +/- 2 weeks, and Month 12 visit occurred 12 months post Day 1 +/- 2 weeks or within 2 weeks after end of treatment. Responder was the participant who achieved TTR stabilization (ie, who had been TTR stabilized). Declaring a participant to have been (TTR) 'stabilized' was defined as the participant whose percent stabilization was equal to or greater than 32%. Percent stabilization (%) was calculated as ([fraction of initial {FOI} dosed - FOI baseline] / FOI baseline)×100, and FOI was calculated as average TTR tetramer concentration (post-denaturation) / average TTR concentration (pre-denaturation).
Time Frame: Predose on Day 1 (baseline), predose and 3 hours post dose at Month 1 visit, 7 hours post dose at Month 6 visit, and 1 hour post dose at Month 12 visit
Population: Pharmacodynamic (PD) analysis set included all enrolled participants who took at least 1 dose of tafamidis free acid 61 mg soft capsule and who had at least 1 TTR stabilization value. Number of Participants Analyzed represents the number of participants who had PD samples collected, and both the baseline and post dose TTR and TTR tetramer concentrations >= the lower limit of quantification (LLOQ). Number Analyzed for each row represents the number of evaluable participants at each timepoint.
Measure: Number (95% Confidence Interval); unit: Percentages of participants
Arm/Group | All Participants
Number analyzed (Participants) | 30
Percentages of participants
  Predose at Month 1: number analyzed (Participants) | 28
  Predose at Month 1 | 96.4 [81.7 to 99.9]
  3 hours post dose at Month 1: number analyzed (Participants) | 28
  3 hours post dose at Month 1 | 96.4 [81.7 to 99.9]
  7 hours post dose at Month 6: number analyzed (Participants) | 26
  7 hours post dose at Month 6 | 96.2 [80.4 to 99.9]
  1 hour post dose at Month 12: number analyzed (Participants) | 19
  1 hour post dose at Month 12 | 94.7 [74.0 to 99.9]

6. Secondary Outcome: TTR Concentration at Baseline, Months 1, 6, and 12
Description: One K2EDTA blood sample of approximate 10 mL was collected on Day 1 (baseline), and at Months 1, 6, and 12 visits for measurement of TTR concentration. Month 1 visit occurred 1 month post Day 1 +/- 1 week, Month 6 visit occurred 6 months post Day 1 +/- 2 weeks, and Month 12 visit occurred 12 months post Day 1 +/- 2 weeks or within 2 weeks after end of treatment.
Time Frame: as for outcome 5
Population: PD analysis set included all enrolled participants who took at least 1 dose of tafamidis free acid 61 mg soft capsule and who had at least 1 TTR concentration value. Number of Participants Analyzed represents the total number of participants in the PD analysis set. Number Analyzed for each row represents the number of participants with evaluable values at the specific timepoints.
Measure: Mean (Standard Deviation); unit: Milligrams per deciliter (mg/dL)
Arm/Group | All Participants
Number analyzed (Participants) | 53
Milligrams per deciliter (mg/dL)
  Predose on Day 1 (baseline) | 12.70 (5.670)
  Predose at Month 1: number analyzed (Participants) | 47
  Predose at Month 1 | 19.73 (7.019)
  3 hours post dose at Month 1: number analyzed (Participants) | 47
  3 hours post dose at Month 1 | 19.58 (6.547)
  7 hours post dose at Month 6: number analyzed (Participants) | 45
  7 hours post dose at Month 6 | 21.48 (7.717)
  1 hour post dose at Month 12: number analyzed (Participants) | 31
  1 hour post dose at Month 12 | 21.79 (7.003)

7. Secondary Outcome: Change From Baseline for Kansas City Cardiomyopathy Questionnaire Overall Summary (KCCQ-OS) Scores at Months 6 and 12
Description: The KCCQ is a self-administered, 23-item questionnaire. KCCQ-OS scores are transformed to a 0 to 100 range, with lower scores denoting poorer quality of life.
Time Frame: Day 1 (baseline), Months 6, and 12
Population: Efficacy analysis set included all enrolled participants who took at least 1 dose of tafamidis free acid 61 mg soft capsule. Number of Participants Analyzed represents the total number of participants in the efficacy analysis set regardless of the type of outcome measures. Number Analyzed for each row represents the number of evaluable participants who had reportable KCCQ-OS scores at baseline, at Months 6 (for reporting CFB at Month 6) and 12 (for reporting CFB at Month 12).
Measure: Mean (Standard Deviation); unit: Score on a scale of 100
Arm/Group | All Participants
Number analyzed (Participants) | 53
Score on a scale of 100
  Month 6: number analyzed (Participants) | 47
  Month 6 | -0.4 (18.97)
  Month 12: number analyzed (Participants) | 43
  Month 12 | -0.3 (19.89)

8. Secondary Outcome: Change From Baseline for EuroQol 5 Dimensions 5 Levels (EQ-5D-5L) Index Values at Months 6 and 12
Description: The EQ-5D-5L is a brief, self-administered generic health status instrument. The instrument consists of 2 parts. In the first part, respondents are asked to rate their current health state on 5 dimensions (mobility, self-care, usual activities, pain or discomfort, and anxiety or depression) with each dimension having 5 levels of function (no problems, slight problems, moderate problems, severe problems, and extreme problems). The second part is a participant's self-rating of current health state on a Visual Analog Scale (EQ-5D VAS) with endpoints labeled 'best imaginable health state' (score of 100) and 'worst imaginable health state' (score of 0). The index values were calculated using the scoring algorithm based on preferences solicited from the Chinese population with 0 representing death and 1 representing full health. Higher EQ-5D-5L index value indicated a better quality of life. Change from baseline for EQ-5D-5L index values are reported for this outcome measure.
Time Frame: Day 1 (baseline), Months 6, and 12
Population: Efficacy analysis set included all enrolled participants who took at least 1 dose of tafamidis free acid 61 mg soft capsule. Number of Participants Analyzed represents the total number of participants in the efficacy analysis set regardless of the type of outcome measures. Number Analyzed for each row represents the number of evaluable participants who had reportable EQ-5D-5L scores at baseline, Months 6 (for reporting CFB at Month 6) and 12 (for reporting CFB at Month 12).
Measure: Mean (Standard Deviation); unit: Index value on a scale of 0-1
Arm/Group | All Participants
Number analyzed (Participants) | 53
Index value on a scale of 0-1
  Month 6: number analyzed (Participants) | 47
  Month 6 | 0.0 (0.24)
  Month 12: number analyzed (Participants) | 43
  Month 12 | 0.0 (0.21)

9. Secondary Outcome: Change From Baseline for EuroQol VAS at Months 6 and 12
Description: The EQ-5D-5L (5 levels version) is a brief, self-administered generic health status instrument. The instrument consists of 2 parts. In the first part, respondents are asked to rate their current health state on 5 dimensions (mobility, self-care, usual activities, pain or discomfort, and anxiety or depression) with each dimension having 3 levels of function (no problems, slight problems, moderate problems, severe problems and extreme problems). The second part is a participant's self-rating of current health state on a EQ-5D VAS with endpoints labeled 'best imaginable health state' (score of 100) and 'worst imaginable health state' (score of 0). The scores from the 5 dimensions may be used to calculate a single index value, also known as a utility score. EQ-5D VAS scores are reported for this outcome measure.
Time Frame: Day 1 (baseline), Months 6, and 12
Population: Efficacy analysis set included all enrolled participants who took at least 1 dose of tafamidis free acid 61 mg soft capsule . Number of Participants Analyzed represents the total number of participants in the efficacy analysis set regardless of the type of outcome measures. Number Analyzed for each row represents the number of evaluable participants who had reportable EuroQol VAS scores at baseline, Months 6 (for reporting CFB at Month 6) and 12 (for reporting CFB at Month 12).
Measure: Mean (Standard Deviation); unit: Score on a scale of 100
Arm/Group | All Participants
Number analyzed (Participants) | 53
Score on a scale of 100
  Month 6: number analyzed (Participants) | 47
  Month 6 | -0.6 (20.23)
  Month 12: number analyzed (Participants) | 43
  Month 12 | 3.4 (15.65)

10. Secondary Outcome: Change From Baseline for Physical Component Summary (PCS) for Short-Form Survey 12 (SF-12) at Months 6 and 12
Description: SF-12 is developed as a shorter alternative to the SF-36 for use in large-scale studies. It is an instrument with different weights for scoring physical and mental health, and measures health-related quality of life with 12 items categorized in eight areas: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health. This questionnaire was completed by the participant after the KCCQ and EQ-5D-5L, and prior to other required visit assessments. PCS score ranges from 0 to 100, and higher PCS score indicates a better quality of life. Change from baseline for PCS for SF-12 is reported for this outcome measure.
Time Frame: Day 1 (baseline), Months 6, and 12
Population: Efficacy analysis set included all enrolled participants who took at least 1 dose of tafamidis free acid 61 mg soft capsule. Number of Participants Analyzed represents the total number of participants in the efficacy analysis set regardless of the type of outcome measures. Number Analyzed for each row represents the number of evaluable participants who had reportable PCS scores at baseline, Months 6 (for reporting CFB at Month 6) and 12 (for reporting CFB at Month 12).
Measure: Mean (Standard Deviation); unit: Score on a scale of 100
Arm/Group | All Participants
Number analyzed (Participants) | 53
Score on a scale of 100
  Month 6: number analyzed (Participants) | 47
  Month 6 | 0.1 (8.24)
  Month 12: number analyzed (Participants) | 43
  Month 12 | -0.0 (9.14)

11. Secondary Outcome: Change From Baseline for Mental Component Summary (MCS) for SF-12 at Months 6 and 12
Description: SF-12 is developed as a shorter alternative to the SF-36 for use in large-scale studies. It is an instrument with different weights for scoring physical and mental health, and measures health-related quality of life with 12 items categorized in eight areas: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health. This questionnaire was completed by the participant after the KCCQ and EQ-5D-5L, and prior to other required visit assessments. MCS score ranges from 0 to 100, and higher MCS score indicates a better quality of life. Change from baseline for MCS for SF-12 is reported for this outcome measure.
Time Frame: Day 1 (baseline), Months 6, and 12
Population: Efficacy analysis set included all enrolled participants who took at least 1 dose of tafamidis free acid 61 mg soft capsule. Number of Participants Analyzed represents the total number of participants in the efficacy analysis set regardless of the type of outcome measures. Number Analyzed for each row represents the number of evaluable participants who had reportable MCS scores at baseline, Months 6 (for reporting CFB at Month 6) and 12 (for reporting CFB at Month 12).
Measure: Mean (Standard Deviation); unit: Score on a scale of 100
Arm/Group | All Participants
Number analyzed (Participants) | 53
Score on a scale of 100
  Month 6: number analyzed (Participants) | 47
  Month 6 | 1.4 (10.60)
  Month 12: number analyzed (Participants) | 43
  Month 12 | 1.5 (12.54)

12. Secondary Outcome: Plasma Concentrations of Tafamidis at Months 1, 6, and 12
Description: Blood samples of approximately 3 mL, to provide an approximately 1 mL plasma, were collected for measurement of plasma concentrations of tafamidis at Months 1, 6, and 12 visits. Month 1 visit occurred 1 month post Day 1 +/- 1 week, Month 6 visit occurred 6 months post Day 1 +/- 2 weeks, and Month 12 visit occurred 12 months post Day 1 +/- 2 weeks or within 2 weeks after end of treatment.
Time Frame: Predose and 3 hours post dose at Month 1 visit, 7 hours post dose at Month 6 visit, and 1 hour post at Month 12 visit
Population: Pharmacokinetic (PK) analysis set included all enrolled participants who took at least 1 dose of tafamidis free acid 61 mg soft capsule and who had at least 1 quantifiable plasma tafamidis concentration. Number of Participants Analyzed represents the number of participants who had at least 1 tafamidis concentration >=LLOQ. Number Analyzed for each row represents the number of participants with non-missing concentrations at each timepoint.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | All Participants
Number analyzed (Participants) | 47
nanograms per milliliter (ng/mL)
  Predose at Month 1 | 10410 (5521.1)
  3 hours post dose at Month 1 | 12040 (4950.1)
  7 hours post dose at Month 6: number analyzed (Participants) | 45
  7 hours post dose at Month 6 | 14100 (5950.5)
  1 hour post dose at Month 12: number analyzed (Participants) | 31
  1 hour post dose at Month 12 | 11950 (5475.8)

ADVERSE EVENTS:
Time Frame: From the first dose of study intervention up to 28 days post the last dose of study intervention (up to a maximum of 393 days)
Description: The same event may appear as both an AE and an SAE. However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as non-serious in another participant, or 1 participant may have experienced both a serious and non-serious event during the study. Total number at risk below refers to the number of participants evaluable for AEs.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 6/53
Serious Adverse Events (participants affected / at risk) | 21/53
Other Adverse Events (participants affected / at risk) | 35/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=53)
Atrial thrombosis (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 6
Cardiac failure acute (Cardiac disorders) | 3
Cardiorenal syndrome (Cardiac disorders) | 1
Hereditary neuropathic amyloidosis (Congenital, familial and genetic disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Disease progression (General disorders) | 2
Oedema peripheral (General disorders) | 1
COVID-19 (Infections and infestations) | 3
Erysipelas (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Respiratory tract infection (Infections and infestations) | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Dizziness (Nervous system disorders) | 1
Haemorrhagic cerebral infarction (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Chronic kidney disease (Renal and urinary disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=53)
Diarrhoea (Gastrointestinal disorders) | 6
Vomiting (Gastrointestinal disorders) | 4
Hepatic function abnormal (Hepatobiliary disorders) | 4
COVID-19 (Infections and infestations) | 12
Nasopharyngitis (Infections and infestations) | 4
Pneumonia (Infections and infestations) | 3
Hyperuricaemia (Metabolism and nutrition disorders) | 5
Haematuria (Renal and urinary disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2021-03-26): https://cdn.clinicaltrials.gov/large-docs/86/NCT04814186/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-07): https://cdn.clinicaltrials.gov/large-docs/86/NCT04814186/SAP_001.pdf